CLINICAL TRIAL: NCT02413138
Title: A Randomized, Phase 2/3, Open-Label, Multi-center Study of the Pharmacokinetics, Pharmacodynamics, Safety and Efficacy of A Long-acting Human Growth Hormone (Somavaratan, VRS-317) in Pre-pubertal Japanese Children With Growth Hormone Deficiency (GHD)
Brief Title: Versartis Trial in Pre-pubertal Japanese Children With Growth Hormone Deficiency (GHD) to Assess Long-Acting Growth Hormone (Somavaratan, VRS-317)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The primary endpoint of non-inferiority to daily therapy in the pediatric Phase 3 study was not achieved
Sponsor: Versartis Inc. (Industry)
Responsible Party: Sponsor
Organization: Aravive, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J14VR5
Record Dates: First submitted 2015-03-23; First posted 2015-04-09 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Pediatric Growth Hormone Deficiency; Growth Disorders
Keywords: GHD
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 2: Somavaratan (VRS-317) (Experimental): Active treatment arm
  Interventions: Drug: Somavaratan (VRS-317)
- Phase 3: Somavaratan (VRS-317) (Experimental): Somavaratan long acting recombinant human growth hormone administered subcutaneously twice-monthly
  Interventions: Drug: Somavaratan (VRS-317)

INTERVENTIONS:
Drug: Somavaratan (VRS-317) — Long acting recombinant human growth hormone
  Other Names: Long acting recombinant human growth hormone

SUMMARY:
The trial will consist of three stages: 1) a 30 day Phase 2 PK and PD evaluation of somavaratan, 2) an optional Phase 2 Extension and 3) a 12 month Phase 3 safety and efficacy stage. Upon completion of the PK/PD stage, the PK/PD profiles for the GHD children in this study will be compared to the PK/PD profiles for the GHD children treated in the Western study Phase 1b/2a study (Protocol 12VR2) and identify the somavaratan dose to be used in the Phase 3 stage in Japan. The Phase 3 stage will continue dosing for 12 months to obtain safety and efficacy data on 48 subjects.

DETAILED DESCRIPTION:
The trial will consist of three stages: 1) a 30 day Phase 2 PK and PD evaluation of somavaratan, 2) an optional Phase 2 Extension and 3) a 12 month Phase 3 safety and efficacy stage. The study is a randomized, multi-center, open label study. The primary endpoint is height velocity at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Chronological Age ≥ 3.0 years and ≤ 9.0 years (girls) or ≤ 10.0 years (boys)
* Pre-pubertal status
* Diagnosis of GHD as documented by two or more GH stimulation test results
* Height SD score ≤ -2.0 at screening
* Weight for Stature ≥ 10th percentile
* IGF-I SD score ≤ -1.0 at screening
* Delayed bone age

Exclusion Criteria:

* Prior treatment with any growth promoting agent
* History of, or current, significant disease
* Chromosomal aneuploidy, significant gene mutations (other than those that cause GHD) or confirmed diagnosis of a named syndrome
* Birth weight and/or birth length less than 5th percentile for gestational age
* A diagnosis of Attention Deficit Hyperactivity Disorder
* Daily use of anti-inflammatory doses of glucocorticoid
* Prior history of leukemia, lymphoma, sarcoma or cancer
* Ocular findings suggestive of increased intracranial pressure and/or retinopathy at screening
* Significant spinal abnormalities including scoliosis, kyphosis and spina bifida variants
* Significant abnormality in screening laboratory studies

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy (Annual Height velocity) | 12 months
  Annual Height velocity.

SECONDARY OUTCOMES:
Pharmacodynamics (IGF-I responses to study drug administration) | 12 months
  IGF-I responses to study drug administration.
Pharmacodynamics (IGFBP-3 responses to study drug administration) | 12 months
  IGFBP-3 responses to study drug administration.
Safety (Number of subjects with adverse events ) | 12 months
  Number of subjects with adverse events (including repeat dose immunogenicity).
Safety (Concomitant medications) | 12 months
  Concomitant medications
Safety (Safety labs) | 12 months
  Safety labs
Safety (Vital signs) | 12 months
  Vital signs
Safety (Physical Exams) | 12 months
  Physical Exams

OTHER OUTCOMES:
Secondary Efficacy (Change in height SDS) | 12 months
  Change in height SDS.
Secondary Efficacy | 12 months
  Change in body weight
Secondary Efficacy | 12 months
  Change in body mass index.
Secondary Efficacy (Change in bone age) | 12 months
  Change in bone age.
Secondary Efficacy (Change in pubertal staging.) | 12 months
  Change in pubertal staging.

CONTACTS AND LOCATIONS:
Overall Officials: Will Charlton, MD, Study Director — Vesrartis
Locations (1):
- Hokkaido University Hospital, Sapporo, Japan

IPD SHARING:
Plan to Share IPD: No